CLINICAL TRIAL: NCT05529693
Title: Efficacy of a Probiotic Strain on Level of Markers of Inflammation in an Elderly Population - a Randomized, Double-blind, Placebo-controlled, Parallel Group Pilot Study With 12 Weeks Intervention
Brief Title: Efficacy of a Probiotic Strain on Level of Markers of Inflammation in an Elderly Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chr Hansen (Industry)
Responsible Party: Sponsor
Organization: ChrHansen (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HND-IM-047
Record Dates: First submitted 2022-08-17; First posted 2022-09-07 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-12

CONDITIONS: Inflammation
MeSH Terms: conditions — Inflammation | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bif-038 arm, high dose (Experimental): Active trial product with minimum 10 billion CFU daily dose
  Interventions: Dietary Supplement: Experimental: Bif-038 arm, high dose
- Bif-038 arm, low dose (Experimental): Active trial product with minimum 1 billion CFU daily dose
  Interventions: Dietary Supplement: Experimental: Bif-038 arm, low dose
- Placebo arm (Placebo Comparator): Similar trial product, but without Bif-038 probiotic bacteria
  Interventions: Dietary Supplement: Placebo Comparator: Placebo arm

INTERVENTIONS:
Dietary Supplement: Experimental: Bif-038 arm, high dose — Active trial product with minimum 10 billion CFU daily dose
  Other Names: Probiotic
  Arms: Bif-038 arm, high dose
Dietary Supplement: Experimental: Bif-038 arm, low dose — Active trial product with minimum 1 billion CFU daily dose
  Other Names: Probiotic
  Arms: Bif-038 arm, low dose
Dietary Supplement: Placebo Comparator: Placebo arm — Similar product to trial product but without Bif-038
  Other Names: Placebo
  Arms: Placebo arm

SUMMARY:
To investigate the effectiveness of two doses of the probiotic strain Bif-038 on markers of low-grade inflammation in a elderly population

DETAILED DESCRIPTION:
The study is a randomized, double-blind, 3-arm, placebo-controlled pilot study in an elderly population (60-85 years) with low-grade inflammation (hs-CRP 2-10 mg/L) comparing two doses daily intake of Bif-038 at 1 and 10 billion CFU to placebo for 12 weeks. The subjects will receive either one of the two test products or the placebo product daily for a period of 12 weeks.

During the entire study period, five visits are scheduled. The subjects will participate in two screening visits; a baseline visit, a visit after 6 weeks of intervention and an end-of-study visit after 12 weeks of intervention. Visit 1 and 2 are screening- and recruitment visits with at least two weeks apart. Only participants with a hs-CRP within 2.0-10.0 mg/L will be invited for the second screening visit. Participants with repeated hs-CRP levels within 2.0-10.0 mg/L will be invited for baseline visit 3, to be included and randomized in the study.

At the screening visits the eligibility will be checked after the participants have given their written informed consent.

Blood samples and stool samples will be collected during the study and subjects will be asked to complete questionnaires and a dietary diary.

No sample size calculations were performed due to the exploratory nature of a pilot study design. Planned number to include is 20 subjects per study arm, thus 60 subjects in total.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate in the study and comply with its procedures
* Able to give written informed consent
* Healthy adults as determined by the investigator
* Age: ≥ 60 years and ≤ 85 years
* hs-CRP: 2.0-10.0 mg/L
* BMI: 18.5-32 kg/m2
* Temperature between ≥35.5 and ≤37.3oC
* A stable body weight (≤5 % change) over the 3 months prior to screening.

Exclusion Criteria:

1. Cold or flu-like (URTI) symptoms, with a Jackson Cold Scale score of >2; not otherwise explained by seasonal allergies
2. Chronic disease such as, cardiovascular diseases, gastrointestinal disorders, and rheumatoid arthritis, which in the Investigators judgment, precludes involvement in the study
3. Oral antibiotics within 4 weeks prior to the screening visit
4. Use of immunosuppressant drugs, systemic steroids or systemic antimicrobial medication (including suppositories) within the 4 weeks prior to the screening visit
5. Regular oral non-steroidal anti-inflammatory medication use (1 week) (topical NSAIDS allowed). Low-dose prophylactic aspirin use is acceptable if stable for 9 months prior to screening.
6. Uncontrolled, unstable hypertension at the discretion of the investigator.
7. Current smoking, chewable tobacco and/or vaping. Low dose (<50mg/week) nicotine products allowed.
8. Planned change in current diet or exercise habits
9. Habitual intake of probiotic supplements within 2 months before screening visit
10. Have had gastrointestinal surgery (e.g. colectomy, cholecystectomy, gastric bypass); Appendectomy allowed. Laparoscopic surgeries (removal of polyps, cysts) are allowed.
11. Have had any other condition or are taking a medication that the investigator believes would interfere with the objectives of the study, pose a safety risk, or confound the interpretation of the study results;
12. Any change in medication or supplement intake in the 30 days prior to baseline
13. Any major dietary changes in the 30 days prior to baseline
14. Has a history of drug and/or alcohol abuse at the time of enrolment;
15. Has received treatment involving experimental drugs in 2 months prior to screening
16. Any immunosuppressant or chemotherapy medications, including marcaptopurine, azothioprine, or methotrexate;
17. Use of herbal remedies and supplements with potential anti-inflammatory properties for the duration of the study, which in the Investigators judgement may have an impact on the objectives of the study.
18. Have a current malignant disease or any current concomitant end-stage organ disease, which, in the Investigator's judgment, contraindicates participation in the study;
19. Individuals who, in the opinion of the investigator, are considered to be poor clinical attendees or unlikely for any reason to be able to comply with the trial.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-09-29 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
hs-CRP | 12 weeks
  The effect of daily intake of Bif-038 10 billion CFU versus placebo on hs-CRP

SECONDARY OUTCOMES:
TNF-alfa | 12 weeks
  The effect of daily intake of Bif-038 10 billion CFU versus placebo on TNF-alfa

OTHER OUTCOMES:
Change in hsCRP | 6 and 12 weeks
  The effect of daily intake of Bif-038 on hsCRP. Comparison between all three treatment groups
Change in TNF-alfa | 6 and 12 weeks
  The effect of daily intake of Bif-038 on TNF-alfa. Comparison between all three treatment groups
Change in feces borne biomarker calprotectin | 12 weeks
  The effect of daily intake of Bif-038 on feces borne biomarker calprotectin. Comparison between all three treatment groups.
Change in Health-related Quality of Life | 6 and 12 weeks
  The effect of daily intake of Bif-038 on changes in heath-related quality of life measured by Short Form 36 questionnaire (SF36). Comparison between all three treatment groups.
  The 36 questions (items) are transformed to 8 dimensions (Physical Functioning, Social Functioning, Role limitations due to physical problems, Role limitations due to emotional problems, Mental health, Energy/vitality, Pain, and General health perception). These 8 dimensions are then again aggregated into two summary scores, physical component and mental health between 0-100 for all dimensions. The lower the score the more disability and the higher the score the less disability.
Change in mental health | 6 and 12 weeks
  The effect of daily intake of Bif-038 on change in mental health measured by Depression Anxiety Scale (DASS-21). Comparison between all three treatment groups.
  The DASS yields three subscale scores for depression, anxiety, and tension/stress. The higher the score the more severe with the following ranging:
  Depression: Normal: 0-9, Mild: 10-12, Moderate:13-20, Severe: 21-27, and Extremely severe: 28-42.
  Anxiety: Normal: 0-6, Mild: 7-9, Moderate: 10-14, Severe:15-19, and Extremely severe: 20-42.
  Stress: Normal: 0-10, Mild:11-18, Moderate:19-26, Severe: 27-34, and Extremely severe: 35-42.
Change in well-being | 6 and 12 weeks
  The effect of daily intake of Bif-038 on change in well-being measured by WHO (Five) Well Being Index. Comparison between all three treatment groups.
  The total raw score, ranging from 0 to 25, is multiplied by 4 to give the final score, with 0 representing the worst imaginable well-being and 100 representing the best imaginable well-being.
Change in microbiome | 12 weeks
  The effect of daily intake of Bif-038 on change in microbiome. Comparison between all three treatment groups
Change in Zonulin | 6 and 12 weeks
  The effect of daily intake of Bif-038 on plasma zonulin. Comparison between all three treatment groups
Change in lipopolysaccharide-binding protein | 6 and 12 weeks
  The effect of daily intake of Bif-038 on plasma lipopolysaccharide-binding protein. Comparison between all three treatment groups
Change in intestinal fatty-acid binding protein | 6 and 12 weeks
  The effect of daily intake of Bif-038 on plasma Intestinal fatty-acid binding protein. Comparison between all three treatment groups
Change in CD4/CD8 ratio | 6 and 12 weeks
  The effect of daily intake of Bif-038 on change in CD4/CD8 ratio. Comparison between all three treatment groups
Change in Interleukin-6 | 6 and 12 weeks
  The effect of daily intake of Bif-038 on serum Interleukin-6. Comparison between all three treatment groups
Change in Interleukin-10 | 6 and 12 weeks
  The effect of daily intake of Bif-038 on serum Interleukin-10. Comparison between all three treatment groups
Change in body weight | 6 and 12 weeks
  The effect of daily intake of Bif-038 on change in body weight. Comparison between all three treatment groups

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Dinan, Professor, Principal Investigator — Atlantia Clinical Trials
Locations (1):
- Atlantia Food Clinical Trials, Cork, Ireland

IPD SHARING:
Plan to Share IPD: No